CLINICAL TRIAL: NCT00707772
Title: A Study on PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin) in Iranian Hemophilic Patients With Chronic Hepatitis C Infection
Brief Title: Pegasys® Plus Ribavirin in Hemophilic Patients With Hepatitis C Virus Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Baqiyatallah Research Center for Gastroenterology and Liver Diseases (Other); Tehran Hepatitis Center (Other); Guilan University of Medical Sciences (Other); Tabriz Research Center for Gastroenterology and Liver Diseases (Unknown); Shahid Beheshti University of Medical Sciences (Other); Iran University of Medical Sciences (Other)
Responsible Party: Professor Seyed-Moayed Alavian, Baqiyatallah Research Center for Gastroenterology and Liver Diseases
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRCGL-07-03; BRCGL-07-03
Record Dates: First submitted 2008-06-26; First posted 2008-07-01 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C; Hemophilia
Keywords: Hepatitis C; Hemophilia; Pegasys; Ribavirin
MeSH Terms: conditions — Hepatitis C; Hemophilia A | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Genotype 2 or 3 in Hemophilic Patients with HCV
  Interventions: Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin)
- 2 (Active Comparator): Other Genotypes (except 2 or 3) in Hemophilic Patients with HCV
  Interventions: Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin)

INTERVENTIONS:
Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin) — PEGASYS: 180 microgram per week (Injection) Plus Ribavirin: 800 milligram per day (PO)
  Other Names: Peginterferon Alfa-2a (40KD) Plus COPEGUS
  Arms: 1
Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin) — PEGASYS: 180 microgram per week (Injection) Plus Ribavirin: [=<75 kg: 1000 mg; >75 kg: 1200 mg per day (PO)]
  Other Names: Peginterferon Alfa-2a (40KD) plus COPEGUS
  Arms: 2

SUMMARY:
Hemophilic patients are a known high risk groups for acquiring the hepatitis C. The surveillance data from Ministry Of Health in IR.Iran had shown that 60% of them are infected with HCV infection. We are trying the PEGASYS plus Ribavirin in Hemophilic patients with HCV.

DETAILED DESCRIPTION:
The investigators enroll 400 patients into the study. The patients receive PEGASYS (Peginterferon alpha-2a(40 KD)) 180 microgram per week plus COPEGUS (Ribavirin) 800 microgram for Genotype 2 and 3 and 1000 milligram for weight less than 75 kg and 1200 milligram for more than 75 kg. The duration of protocol is depends on genotypes of virus. In genotype 1 and 4, for 48 week and in genotypes 2 and 3 , for 24 weeks. The patients are visited every 4 weeks with biochemistry lab tests. The patients are checked with quantitative HCV RNA on the third months after initiation of the treatment to assess early virologic response and at the end of the study for complete response rate and on the six month after treatment completion for sustained response rate. The patients with undetectable HCV RNA are considered as responders. We have omitted the liver biopsy in the patients.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive
* Age older than 12 years

Exclusion Criteria:

* Ongoing pregnancy or breast feeding
* Hx of HCC
* Hx of alcoholic liver disease
* Hx of bleeding from esophageal varices
* Hx of hemochromatosis
* Hx of autoimmune hepatitis
* Hx of Suicidal attempt
* Hx of cerebrovascular dis
* Hx of severe retinopathy
* Hx of severe psoriasis
* Hx of scleroderma
* Hx of metabolic liver disease
* Hx of SLE

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Early Virologic Response | After 12 weeks of Treatment
End of Treatment Response | 24 weeks for : Genotype 2 & 3; 48 Weeks for other genotype
Sustained Virologic Response | 24 weeks after Treatment
Rapid Virologic Response | One month after Treatment

SECONDARY OUTCOMES:
Tolerability of drugs for whole therapy period | During Treatment
Biochemical response (ALT) | End of Treatment AND 24 weeks after Treatment
Laboratory Parameters | During Treatment AND End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Seyed-Moayed Alavian, Professor, Study Chair — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Seyyed Mohammad Miri, M.D., Study Director — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Maryam Keshvari, M.D., Principal Investigator — Iranian blood Transfusion Research Center; Bita Behnava, M.D., Principal Investigator — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Mohammad Hossein Somi, M.D., Principal Investigator — Research Center for Gastroenterology and Hepatology, Tabriz University of Medical Sciences, Tabriz; Fariborz Mansour-Ghanaei, M.D., Principal Investigator — Gastroenterology and Liver Diseases, Gastrointestinal and Liver Diseases Research Center (GLDRC), Guilan University of Medical Sciences, Rasht, Iran; Pegah Karimi, M.D., Principal Investigator — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Bashir HajiBeigi, M.D., Principal Investigator — Iranian Blood Transfusion Research Center
Locations (1):
- Baqiyatallah Research Center for Gastroenterology and Liver Diseases, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Iafolla M. [Pegasys: FDA approved Pegasys (peginterferon alfa-2a) for the treatment of hepatitis C]. Sidahora. 2002;(4):8-10. No abstract available. Spanish. PMID 12703472